CLINICAL TRIAL: NCT00073060
Title: Citrate Effects and Bone Density Studies in Long-Term Apheresis Donors
Brief Title: Citrate Effects and Bone Density in Long-Term Apheresis Donors
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 040046; 04-CC-0046
Record Dates: First submitted 2003-11-14; First posted 2003-11-17 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Healthy Apheresis Donors
Keywords: Hypocalcemia; Plateletpheresis; Calcium; Citrate; Bone Density; Natural History; Healthy Volunteer; HV
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NIH Platelepheresis Donors: 75, Apheresis Study Group - donation procedures use same devices as leukapheresis donors, also requiring citrate infusion
- NIH Research Leukapheresis Donors: 75, Apheresis Study Group - donation procedures use same devices as plateletpheresis donors, also requiring citrate infusion; citrate administered may be twice as great as during plateletpheresis.
- NIH Whole Blood Donors: 150 age, gender, race-matched donors - CONTROL GROUP

SUMMARY:
This study will examine the effects of repeated apheresis procedures on bone density and calcium balance. Apheresis is a procedure for collecting large numbers of a specific blood component, such as white cells (leukapheresis) or platelets (plateletpheresis). For the procedure, whole blood is collected through a needle in an arm vein and is directed through a machine that separates it into its components by spinning. The desired cells are removed and the rest of the blood is returned to the donor, either through the same needle or through a needle in the other arm. A blood thinning medicine called citrate is added to the cell-separating machine. Citrate reduces the ionized calcium levels in the blood, which prevents the blood from clotting. When the blood is returned to the donor, the donor also receives the citrate. This lowers the donor's ionized calcium levels which may irritate nerve and muscle cells, causing tingling around the mouth, hands, and feet during the procedure. The reduced ionized calcium levels result in increased parathyroid hormone levels in the donor, can effect bone calcium stores. In addition, some of the citrate that is returned to the donor is excreted in the urine along with calcium, which causes further loss of calcium from the body. It is not known if the calcium loss during apheresis in people who undergo this procedure repeatedly has any long-term effects on body calcium balance and bone calcium stores. This study will measure bone density and calcium balance in long-term platelet and white cell donors and compare the findings with those of whole blood donors, who do not receive citrate.

Healthy people between 18 and 80 years of age who weigh between 110 and 300 pounds, do not have a metal prosthesis, and are not pregnant may be eligible for this study. Participants undergo the following procedures:

Whole blood donors

* Blood sample collection 2 weeks before blood donation.
* I removed undergo standard whole blood donation
* Urine sample collection.
* DEXA scan to assess bone density by measuring bone calcium stores. For this procedure, the subject lies still on a table while the spine, hip, and whole body are scanned using a small amount of radiation. The forearm is also scanned while the subject is seated. The scan may be repeated after 2 years.

Plateletpheresis and leukapheresis donors

* Standard platelet or white cell donation.
* Blood sample collections immediately prior to and after donation, and on the first, fourth, and fourteenth days after donation.
* Urine sample collections at the beginning and at the end of the apheresis procedure and on the first, fourth, and fourteenth days after the donation.
* DEXA scan at the beginning of the study (no earlier than 2 weeks after their latest apheresis donation). The scan may be repeated after 2 years.
* Some apheresis donors may be asked to have a second procedure in which they take calcium according to standard guidelines for plateletpheresis and leukapheresis. During the second procedure, platelet donors will take oral calcium tablets before starting plateletpheresis. White cell donors will receive calcium intravenously (through a vein) during the second leukapheresis. For this second procedure, the donors provide additional blood and urine samples as described above.

DETAILED DESCRIPTION:
Approximately one million plateletpheresis procedures are performed each year in the U.S., including 3,500 in the Platelet Center of the Department of Transfusion Medicine, NIH. Healthy donors are eligible to undergo plateletpheresis as often as 24 times per year. During plateletpheresis, citrate anticoagulant is added to the blood collection pathway to prevent clotting in the apheresis device, and is infused into the donor during the procedure.1-3 Adverse effects related to citrate administration are common; the most well-studied is acute hypocalcemia due to the formation of calcium-citrate complexes. Recent studies in our Department indicate that changes in serum calcium, PTH, osteocalcin, alkaline phosphatase, and vitamin D levels are also present and may be sustained for up to 24 hours after apheresis. Observations from European studies suggest that serial plateletpheresis donation may be associated with reduced bone density; however, those studies did not include a control group, and involved paid donors, who generally were generally younger, allowed to donate more frequently, and not representative of the population demographics of the U.S. In addition to volunteer plateletpheresis donors, the NIH Department of Transfusion Medicine maintains a registry of approximately 500 persons who undergo leukapheresis procedures to provide components for in vitro research use, for which they receive compensation. These research apheresis procedures use the same devices as plateletpheresis donations, and also require citrate anticoagulant infusions. However, the procedure duration and total dose of citrate administered may be twice as great as that which occurs during plateletpheresis. Leukocyte and plateletpheresis donors may undergo more than 100 apheresis procedures during the course of their participation in the donor program at NIH. The impact of serial, frequent, long-term apheresis donations on total body calcium balance and bone density are unknown. In this study, we will measure bone density and laboratory tests in 75 NIH plateletpheresis donors, 75 NIH research leukapheresis donors, and in a control group of 150 age, gender, and race matched NIH whole blood donors. The apheresis study groups will each include at least 50 frequent donors (greater than 50 donations during the past 10 years) and 20 donors with less than 25 lifetime donations. Comprehensive laboratory evaluations of the effect of citrate administration on bone metabolism and body calcium and magnesium metabolism before and after apheresis will be performed. Similar laboratory and bone density measurements will be performed in 75 subjects who donate platelets at facilities outside of NIH (non-NIH donors), and who undergo plateletpheresis at more frequent intervals than NIH donors. The effect of intravenous calcium administration on apheresis-induced changes in these laboratory parameters will also be assessed. This information will have a major impact on our understanding of the short and long-term adverse effects of citrate administration in committed apheresis donors, and may also provide insight into calcium, magnesium, and phosphorus metabolism.

ELIGIBILITY:
* INCLUSION CRITERIA:

<TAB>

Healthy donors who meet all American Association of Blood Banks, Food and Drug Administration and NIH DTM criteria for allogeneic or research blood donation and who have donated blood or apheresis components greater than 50 times in the past 10 years period (NIH donors), greater than 100 times in the past 10 years (non-NIH donors), or less than 25 times in their life (NIH donors).

Age greater than or equal to 18 years and less than or equal to 80 years.

Weight greater than or equal to 50 kg and less than 135 kg.

<TAB>

Able to give informed consent

Able to donate as early as 08:00 in the morning (apheresis donors only).

EXCLUSION CRITERIA:

Pregnancy

Metal prosthesis in place

<TAB>

Any prior radiologic contrast administration within preceding one week (includes CT contrast, MRI contrast, intravenous pyelogram, barium swallow or fluoroscopy)

Weight less less than 50 Kg (minimum weight to donate platelets, leukocytes, whole blood)

Weight greater than135 Kg (maximum weight for DEXA Scan)

More than 2 lifetime apheresis donations for whole blood donors (most recent apheresis must be at least one month prior to this study).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing NIH donors@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2003-11-17 (Actual); Primary Completion 2008-08-26 (Actual); Study Completion 2008-08-26 (Actual)

PRIMARY OUTCOMES:
Citrate Effets on Bone Density | Pre & Post Apheresis
  Determine bone density measurements in serial plateletpheresis and leukapheresis donors & compare them to bone density measurements in a control group.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard N Chen, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-CC-0046.html